CLINICAL TRIAL: NCT06383702
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Controlled, Phase 3 Trial to Evaluate the Efficacy and Safety of Pregabalin Sustained-Release Tablets for the Treatment of Neuropathic Pain Associated With Diabetic Peripheral Neuropathy
Brief Title: A Study to Evaluate Pregabalin in Painful Diabetic Peripheral Neuropathy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HEX1939-002
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Painful Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: Parallel design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: pregabalin sustained-release tablets (Experimental)
  Interventions: Drug: pregabalin sustained-release tablets
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pregabalin sustained-release tablets — Subjects will take pregabalin sustained-release tablets for the duration of 14 weeks. The dosage will include 165 mg daily (for the titration and the withdraw period) and 330 mg daily for the fixed-dose period.
  Arms: Experimental: pregabalin sustained-release tablets
Drug: Placebo — Subjects will take placebo tablets for the duration of 14 weeks. The dosage will include 165 mg daily (for the titration and the withdraw period) and 330 mg daily for the fixed-dose period.
  Arms: Placebo Comparator

SUMMARY:
This study is designed to evaluate the efficacy and safety of pregabalin extended-release tablets in the treatment of neuropathic pain associated with diabetic peripheral neuropathy. Pregabalin has been approved in more than 130 countries for neuropathic pain associated with diabetic peripheral neuropathy, postherpetic neuralgia, and neuralgia associated with spinal cord injury. Pregabalin extended-release tablets were administered once daily, as a single dose after dinner. Compared with pregabalin capsule formulation, it reduces the frequency of medication and improves patient compliance.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled trial, the study was designed to evaluate the efficacy and safety of pregabalin sustained-release tablets in the treatment of neuropathic pain associated with diabetic peripheral neuropathy. The study includes a screening period (3 weeks, including baseline/run-in period), a treatment period (titration period, fixed dose period and withdrawal period), and a follow-up period. During the treatment period participants will receive pregabalin sustained-release tablets/placebo as daily treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years and ≤ 75 years at screening;
* diagnosed with type 1 or type 2 diabetes for ≥ 1 year;
* diagnosed with distal symmetrical polyneuropathy caused by diabetes (type 1 or type 2), with duration of neuropathic pain associated with diabetic peripheral neuropathy ≥ 6 months;
* clearly understood and voluntarily participated in the study, and signed the informed consent form by themselves.

Exclusion Criteria:

* Subjects with other conditions that may confound the assessment of Neuropathic Pain associated with Diabetic Peripheral neuropathy (DPNP), such as: neuropathic pain other than DPNP (cervical spondylosis, carpal tunnel syndrome, spinal stenosis, postherpetic pain, etc.), pain caused by other causes (gout, chronic obstructive arteriosclerosis, arthritis, etc.), and other pain at the assessment site (skin diseases and trauma);
* subjects with known or suspected allergic reactions to various components of pregabalin sustained-release tablets or compounds closely related to paracetamol or paracetamol;
* subjects with clinically significant or unstable diseases, such as but not limited to severe cardiovascular disease, cerebrovascular disease, liver, kidney, respiratory system, blood system, immune system diseases, inflammatory or rheumatic diseases, uncontrolled infection, untreated endocrine diseases, etc., and other conditions that judged by the investigator to influence participation in the trial;
* subjects who have undergone renal transplantation, or are undergoing renal dialysis;
* subjects with uncontrolled narrow-angle glaucoma, uncontrolled seizure history, or uncontrolled or poorly controlled hypertension;
* Pregnant or lactating females or subjects planning to father a child during the trial (including males);
* subjects with a history of drug or alcohol abuse within one year prior to screening; patients who, in the opinion of the investigator, are not suitable for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) mean change at week 13. | Week 13
  The NRS is an 11-point scale ranging from zero ("no pain") to ten ("pain as bad as you can imagine") for self-reporting of pain by patients. Change from baseline in weekly mean of NRS (numeric rating scale) at week 13 will be recorded

SECONDARY OUTCOMES:
NRS mean change at Weeks 1-12 and 14 | Weeks 1-12 and 14
  The NRS is an 11-point scale ranging from zero ("no pain") to ten ("pain as bad as you can imagine") for self-reporting of pain by patients. Change from baseline in weekly mean NRS pain score at Weeks 1-12 and 14 during the treatment period will be recorded;
Proportion of subjects with NRS change | Week 13
  The NRS is an 11-point scale ranging from zero ("no pain") to ten ("pain as bad as you can imagine") for self-reporting of pain by patients. Proportion of subjects with ≥ 50% and ≥ 30% change from baseline in weekly mean NRS pain score at Week 13 will be recorded;
Brief McGill Pain Questionnaire (SF-MPQ) score | Weeks 1, 5, 9, 13, and 14
  It is a self-report questionnaire that allows individuals to give their doctor a good description of the quality and intensity of pain that they are experiencing. Users first select a single word from each group that best reflects their pain; then respondents specify their level of pain by indicating a position along a continuous line between two end-points; then subjects chose the numer best represent their current pain intensity (0~5). Change from baseline in SF-MPQ (Brief McGill Pain Questionnaire) total score and each subscale Pain Grading Index (PRI), Visual Analogue Scale (VAS), and Present Pain Intensity (PPI) scores at Weeks 1, 5, 9, 13, and 14 after treatment;
Medical Outcomes Study Sleep Scale (MOS-SS) score | Weeks 1, 5, 9, 13, and 14
  Participants answered a series of 12 questions assessing sleep, with values ranging from 1 to 6, and an additional dichotomous indicator of optimal sleep. All items are scored so that a high score reflects more of the attribute implied by the scale name. Each item is then converted to a 0 to 100 possible range so that the lowest and highest possible scores are set at 0 and 100, respectively. In this format, scores represent the achieved percentage of the total possible score. Change from baseline in MOS-SS sleep scale score and each subscale (sleep interference, sleep adequacy, daytime mental status, snoring, shortness of breath upon awakening, and sleep volume) score at Weeks 1, 5, 9, 13, and 14 after treatment;
Hospital Anxiety and Depression Scale (HADS) score | Weeks 1, 5, 9, 13, and 14
  The HADS is a fourteen-item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. Change from baseline in HADS (Hospital Anxiety and Depression Scale) score at Weeks 1, 5, 9, 13, and 14 after treatment;
Patient Global Impression of Improvement (PGIC) score | Weeks 1, 5, 9, 13, and 14
  The Patient Global Impression of Change (PGIC) is a patient-reported instrument that measures change in overall status on a scale ranging from one ("very much improved") to seven ("very much worse"). The PGIC is based on the validated Clinical Global Impression of Change scale. Change from baseline in PGIC (Patient Global Impression of Improvement) score at Weeks 1, 5, 9, 13, 14 after treatment will be recorded;
Clinical Global Impression of Improvement (CGIC) score | Weeks 1, 5, 9, 13, and 14
  The Clinical Global Impression of Change (PGIC) is a clinician-reported instrument that measures change in overall status on a scale ranging from one ("very much improved") to seven ("very much worse"). Change from baseline in CGIC (Clinical Global Impression of Improvement) score at Weeks 1, 5, 9, 13, 14 after treatment;